CLINICAL TRIAL: NCT02639364
Title: the Effects and Safety of the Early Application of Bi-level Airway Pressure Ventilation-airway Pressure Release Ventilation(BILEVEL-APRV) Protocol and Conventional Ventilation Strategy Were Compared in ARDS Patients
Brief Title: Airway Pressure Release Ventilation (APRV) Protocol Early Used in Acute Respiratory Distress Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Zhou Yongfang, Principal Investigator, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015 approval (156)
Record Dates: First submitted 2015-12-13; First posted 2015-12-24 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-12

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional ventilation strategy (Active Comparator): The conventional ventilation strategy use volume-controlled ventilation (VCV) or pressure-controlled ventilation (PCV) mode, combination with low tidal volume and adequate PEEP level.
  Interventions: Device: Nellcor Puritan Bennett 840 ventilator system
- BILEVEL-APRV protocol (Experimental): According to our BILEVEL-APRV protocol, BILEVEL-APRV APRV mode with specific settings,combination with spontaneous breathing.
  Interventions: Device: Nellcor Puritan Bennett 840 ventilator system

INTERVENTIONS:
Device: Nellcor Puritan Bennett 840 ventilator system — Puritan Bennett 840 ventilator can provide the VCV,PCV,Bi-level Airway Pressure Ventilation-airway Pressure Release Ventilation(BILEVER-APRV) mode.

SUMMARY:
The aim of this study is to assess the effects and safety of the early application of BILEVEL-APRV protocol and conventional ventilation strategy that used low tidal volume and adequate PEEP level in ARDS patients .

DETAILED DESCRIPTION:
Although mechanical ventilation is life-sustaining for patients with ARDS, it can perpetuate lung injury. A number of recent advances have greatly improved in the mechanical ventilation strategies and treatment for acute respiratory distress syndrome (ARDS), however, Mortality remains high, even with the use of low tidal volume and adequate positive end expiratory pressure(PEEP). Numerous experimental showed that the BILEVEL-APRV mode used in animal ARDS model can improve gas exchanges and hemodynamic tolerance of the ventilation while reducing the dosage for sedative drugs.

The aim of this single-center, prospective, randomized, controlled, open study is to compare the effects and safety of the early application of BILEVEL-APRV protocol and conventional ventilation strategy that used low tidal volume and adequate PEEP level in ARDS patients .

ELIGIBILITY:
Inclusion Criteria:

* Acute respiratory distress syndrome,according to the Berlin definition of ARDS, - The receipt of endotracheal mechanical ventilation for a period was no longer than 48 hours
* A ratio of the partial pressure of arterial oxygen (PaO2) to the fraction of inspired oxygen(FiO2) was less than 250.

Exclusion Criteria:

* Pregnancy
* The expected duration of mechanical ventilation was less than 48 hours
* Intracranial hypertension (suspected or confirmed)
* Neuromuscular disorders that are known to prolong the need for mechanical ventilation
* Known or suspected chronic obstructive pulmonary disease(COPD)
* Preexisting conditions with an expected 6-month mortality exceeding 50%
* Pneumothorax (drained or not)at enrollment
* Treatment with extracorporeal support (ECMO) at enrollment
* There was a lack of commitment to life support.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Mechanical ventilation free days | day 28

SECONDARY OUTCOMES:
all causes mortality | day 60
  Participants will be followed for the duration of ICU stay
all cause hospital mortality | day 60
  Participants will be followed for the duration of hospital stay, until day 60 maximum.
Duration of stay in ICU | day 60
Duration of hospital stay | day 60
peak airway pressure,mean airway pressure,positive end expiratory pressure(cmH2O) | day 7
Average dosage of sedative infusion | day 7
Richmond Sedation-Agitation Scale | day 7
Average dosage of vasoactive drugs each day in use | day 7
number of patients requiring cointerventions and Adjunctive Therapies | Day 28
number of patients requiring the use of noninvasive ventilation | Day 28
the tracheotomy rate | Day 28
Number of patients with a pneumothorax | Day 28
the number of days free from organ dysfunction | Day 28
tidal volume(ml) | Day 7
static lung compliance（ml/cmH2O） | Day 7
PaO2,PaCO2(mmHg) | Day 7
Blood pressure(mmHg) | Day 7
blood lactic acid（mmol/l） | Day 7
minute ventilation (L) | Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Yan Kang, doctor, Study Director — West China Hospital
Locations (1):
- Department of Critical care medicine of West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No